CLINICAL TRIAL: NCT02823925
Title: Bisphosphonates in Multicentric Osteolysis, Nodulosis and Arthropathy (MONA) Spectrum Disorder - an Alternative Therapeutic Approach
Brief Title: Bisphosphonate Therapy in MONA Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Karin Pichler, MD PhD, Medical University Innsbruck
Other Study IDs: SREP-16-11962A
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Bone Density; Pain; Fracture
MeSH Terms: conditions — Pain; Fractures, Bone | interventions — Pamidronate; Zoledronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Pamidronate or Zoledronate

SUMMARY:
Multicentric osteolysis, nodulosis and arthropathy (MONA) spectrum disorder is a rare inherited progressive skeletal disorder caused by mutations in the matrix metalloproteinase 2 (MMP2) gene. Treatment options are limited. The investigators reviewed the outcome of patients affected with MONA and treated with intravenous bisphosphonates in the clinical Center.

DETAILED DESCRIPTION:
Assessment of the patients:

After informed consent had been obtained from the patients affected from MONA spectrum disorder the investigators assessed the patients regarding the following characteristics: consanguinity, clinical symptoms at diseases on-set, age at on-set of symptoms and age at diagnosis, cognitive development, progression of clinical symptoms related to the diagnosis, molecular investigations, associated disorders as well as therapies besides bisphosphonate therapy. Informed consent from the patients was also obtained to publish the patient's photographs. All investigations are performed according to the relevant ethical guidelines.

Bisphosphonate therapy:

The reported patients received intravenous bisphosphonate therapy either with pamidronate (1 mg/kg/d on two consecutive days every 3 months) or zoledronate (a single dose of 0.05 mg/kg/day every 6 month).

Evaluation of disease progression and therapeutic success:

To assess both progression of MONA spectrum disorder and therapeutic success the patients were regularly evaluated clinically in 3 to 6 month intervals. Clinical evaluation comprised an internal, neurological and orthopaedic status as well as a general assessment of neurocognitive function. Additionally, need for oral analgesic therapy was documented. In irregular intervals, depending also on the clinical symptoms, x-rays of hand and feet were taken and a densitometry of the total body, lumbar spine and hip was performed.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed MONA spectrum disorder
* treatment with bisphosphonates intravenously
* positive informed consent

Exclusion Criteria:

* genetically confirmed MONA spectrum disorder treated otherwise than with bisphosphonates
* oral treatment with bisphosphonates in MONA spectrum disorder
* other inherited osteolysis syndromes than MONA spectrum disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three siblings were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
bone mineral density | 10 years